CLINICAL TRIAL: NCT02129530
Title: Effect of Community Social Mobilization for the Prevention of HIV in Young South African Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Witwatersrand, South Africa (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Audrey Pettifor, PhD, Principal Investigator, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11-2062
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2016-01-06 (Estimated); Status verified 2016-01

CONDITIONS: Gender Relations
Keywords: Community Mobilization; HIV; Intimate Partner Violence; Gender Norms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community Social Mobilization Program (Experimental): A manualized intervention developed with Sonke Gender Justice Network using a workshop intervention manual and a community mobilization toolkit will be used.
  Interventions: Behavioral: Community Social Mobilization program
- Control Arm (No Intervention): The Control Arm does not receive the Community Mobilization Intervention

INTERVENTIONS:
Behavioral: Community Social Mobilization program
  Arms: Community Social Mobilization Program

SUMMARY:
The overall purpose is to assess whether a community social mobilization (CSM) program focused on young men ages 18-35 years of age changes gender norms in the community. The secondary purpose is to determine if there is a combined effect of CSM and HPTN 068 (Conditional Cash Transfers) on HIV and HSV-2 incidence. The goal of the mobilization activities is to engage young men around the issues of gender norms, intimate partner violence and HIV risk and to encourage them to take action to protect young women and reduce HIV risk in their communities.

ELIGIBILITY:
Inclusion Criteria:

Quantitative Work

* Men and women ages 18-35 years
* Have lived in study area continuously for the past 12 months
* Able and willing to provide informed consent

Qualitative Work

* Men and women ages 18-99 years
* A community member, CAT member or community mobilizer
* Able and willing to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2502 (Actual)
Dates: Start 2012-03; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Changes in Gender Equitable Mens Scale (GEMS) | Baseline and 24 months

SECONDARY OUTCOMES:
The number of unprotected sex acts | Baseline and 24 months
Concurrency | Baseline and 24 months
  The investigators will measure concurrency by assessing the date of first and last sex and whether a relationship is ongoing among the last 3 partners in the last 12 months.
Experience of perpetration of Intimate partner violence (IPV) | Baseline and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Pettifor, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- MRC/WITS and Agincourt Rural Health Transition Research Unit, Bosbokrand, Mpumalanga, South Africa

REFERENCES:
- [Derived] Pettifor A, Lippman SA, Gottert A, Suchindran CM, Selin A, Peacock D, Maman S, Rebombo D, Twine R, Gomez-Olive FX, Tollman S, Kahn K, MacPhail C. Community mobilization to modify harmful gender norms and reduce HIV risk: results from a community cluster randomized trial in South Africa. J Int AIDS Soc. 2018 Jul;21(7):e25134. doi: 10.1002/jia2.25134. PMID 29972287
- [Derived] Pettifor A, Lippman SA, Selin AM, Peacock D, Gottert A, Maman S, Rebombo D, Suchindran CM, Twine R, Lancaster K, Daniel T, Gomez-Olive FX, Kahn K, MacPhail C. A cluster randomized-controlled trial of a community mobilization intervention to change gender norms and reduce HIV risk in rural South Africa: study design and intervention. BMC Public Health. 2015 Aug 6;15:752. doi: 10.1186/s12889-015-2048-z. PMID 26245910